CLINICAL TRIAL: NCT00560118
Title: Phase II Study of the Predictive Value of the Expression of Tumoral MGMT With Respect to the Therapeutic Response of Fotemustine in Patients With Metastatic Malignant Melanoma
Brief Title: Fotemustine in Treating Patients With Metastatic Melanoma
Acronym: MGFOT1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In view of the slowness of the inclusions and the difficulty of carrying out the study, it was decided to put an end to this study.
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574147; RECF0287 (Registry Identifier: INCA)
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — fotemustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Fotemustine (Experimental): Induction treatment Fotémustine 100mg / m² IV sur 1 h J1, J8, J15
  Traitement d'entretien : Fotémustine 100 mg / m² IV sur 1 h - J1 = J21
  Interventions: Drug: fotemustine

INTERVENTIONS:
Drug: fotemustine
  Other Names: experimental arm

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fotemustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors predict how well patients will respond to treatment.

PURPOSE: This phase II trial is studying fotemustine to see how well it works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the relationship between MGMT expression and response to fotemustine in patients with metastatic malignant melanoma.

Secondary

* Establish a value for MGMT expression below which fotemustine has a strong probability of effectiveness.

OUTLINE: This is a multicenter study.

Patients receive induction chemotherapy comprising fotemustine IV over 1 hour on days 1, 8, and 15. Beginning 5 weeks later, patients achieving stable or objective response receive maintenance chemotherapy comprising fotemustine IV over 1 hour once every 3 weeks for 6 courses.

Tissue samples are collected at baseline to assess level of MGMT expression by PCR.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic malignant melanoma, meeting the following criteria:

  * Metastatic lymph nodes or skin allowing for surgical resection
  * At least 1 metastatic lesion (lymph nodes, skin, visceral, brain)
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC > 2 x 10^9/L
* Platelet count > 100 x 10^9/L
* Transaminases ≤ 2.5 times normal
* Alkaline phosphate ≤ 2.5 times normal
* Total bilirubin normal
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No severe uncontrolled infection
* No other prior or concurrent malignancy (except basal cell or squamous cell carcinoma in situ of the cervix that was curatively treated)

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* At least 2 weeks since prior adjuvant therapy
* At least 4 weeks since prior radiotherapy
* At least 30 days since prior participation in another clinical trial
* No prior or concurrent prophylactic phenytoin

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-08-08 (Actual); Primary Completion 2008-08-31 (Actual); Study Completion 2008-08-31 (Actual)

PRIMARY OUTCOMES:
Relationship between MGMT expression and response to fotemustine | from date of inclusion to death of patient
  response with criteria OMS
Relationship between MGMT expression and response to fotemustine | from date of inclusion to progression documentation
  response with criteria OMS

CONTACTS AND LOCATIONS:
Overall Officials: Didier Cupissol, MD, PhD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baughan CA, Hall VL, Leppard BJ, Perkins PJ. Follow-up in stage I cutaneous malignant melanoma: an audit. Clin Oncol (R Coll Radiol). 1993;5(3):174-80. doi: 10.1016/s0936-6555(05)80321-8. PMID 8347541
- [Background] Sirott MN, Bajorin DF, Wong GY, Tao Y, Chapman PB, Templeton MA, Houghton AN. Prognostic factors in patients with metastatic malignant melanoma. A multivariate analysis. Cancer. 1993 Nov 15;72(10):3091-8. doi: 10.1002/1097-0142(19931115)72:103.0.co;2-v. PMID 8221576
- [Background] Battayani Z, Grob JJ, Xerri L, Noe C, Zarour H, Houvaeneghel G, Delpero JR, Birmbaum D, Hassoun J, Bonerandi JJ. Polymerase chain reaction detection of circulating melanocytes as a prognostic marker in patients with melanoma. Arch Dermatol. 1995 Apr;131(4):443-7. PMID 7726587
- [Background] Hauschild A, Michaelsen J, Brenner W, Rudolph P, Glaser R, Henze E, Christophers E. Prognostic significance of serum S100B detection compared with routine blood parameters in advanced metastatic melanoma patients. Melanoma Res. 1999 Apr;9(2):155-61. doi: 10.1097/00008390-199904000-00008. PMID 10380938
- [Background] Kageshita T, Yoshii A, Kimura T, Kuriya N, Ono T, Tsujisaki M, Imai K, Ferrone S. Clinical relevance of ICAM-1 expression in primary lesions and serum of patients with malignant melanoma. Cancer Res. 1993 Oct 15;53(20):4927-32. PMID 8104688
- [Background] Luca M, Hunt B, Bucana CD, Johnson JP, Fidler IJ, Bar-Eli M. Direct correlation between MUC18 expression and metastatic potential of human melanoma cells. Melanoma Res. 1993 Feb;3(1):35-41. doi: 10.1097/00008390-199304000-00006. PMID 8471835
- [Background] Hieken TJ, Ronan SG, Farolan M, Shilkaitis AL, Das Gupta TK. Molecular prognostic markers in intermediate-thickness cutaneous malignant melanoma. Cancer. 1999 Jan 15;85(2):375-82. doi: 10.1002/(sici)1097-0142(19990115)85:23.0.co;2-1. PMID 10023705
- [Background] Smolle J, Hofmann-Wellenhof R, Kerl H. Prognostic significance of proliferation and motility in primary malignant melanoma of the skin. J Cutan Pathol. 1992 Apr;19(2):110-5. doi: 10.1111/j.1600-0560.1992.tb01351.x. PMID 1597566
- [Background] Middleton MR, Grob JJ, Aaronson N, Fierlbeck G, Tilgen W, Seiter S, Gore M, Aamdal S, Cebon J, Coates A, Dreno B, Henz M, Schadendorf D, Kapp A, Weiss J, Fraass U, Statkevich P, Muller M, Thatcher N. Randomized phase III study of temozolomide versus dacarbazine in the treatment of patients with advanced metastatic malignant melanoma. J Clin Oncol. 2000 Jan;18(1):158-66. doi: 10.1200/JCO.2000.18.1.158. PMID 10623706
- [Background] Avril MF, Bonneterre J, Delaunay M, Grosshans E, Fumoleua P, Israel L, Bugat R, Namer M, Cupissol D, Kerbrat P, et al. Combination chemotherapy of dacarbazine and fotemustine in disseminated malignant melanoma. Experience of the French Study Group. Cancer Chemother Pharmacol. 1990;27(2):81-4. doi: 10.1007/BF00689087. PMID 2249337
- [Background] Avril MF, Bonneterre J, Cupissol D, Grob JJ, Kalis B, Fumoleau P, Kerbrat P, Israel L, Fargeot P, Lambert D, et al. Fotemustine plus dacarbazine for malignant melanoma. Eur J Cancer. 1992;28A(11):1807-11. doi: 10.1016/0959-8049(92)90008-p. PMID 1389514
- [Background] Mechl Z, Krejci P. Cis-diamminedichloroplatinum in the treatment of disseminated malignant melanoma. Neoplasma. 1983;30(3):371-7. PMID 6683360
- [Background] Flaherty LE. Rationale for intergroup trial E-3695 comparing concurrent biochemotherapy with cisplatin, vinblastine, and DTIC alone in patients with metastatic melanoma. Cancer J Sci Am. 2000 Feb;6 Suppl 1:S15-20. PMID 10685653
- [Background] Jacquillat C, Khayat D, Banzet P, Weil M, Fumoleau P, Avril MF, Namer M, Bonneterre J, Kerbrat P, Bonerandi JJ, et al. Final report of the French multicenter phase II study of the nitrosourea fotemustine in 153 evaluable patients with disseminated malignant melanoma including patients with cerebral metastases. Cancer. 1990 Nov 1;66(9):1873-8. doi: 10.1002/1097-0142(19901101)66:93.0.co;2-5. PMID 2224783
- [Background] Jacquillat C, Khayat D, Banzet P, Weil M, Avril MF, Fumoleau P, Namer M, Bonneterre J, Kerbrat P, Bonerandi JJ, et al. Chemotherapy by fotemustine in cerebral metastases of disseminated malignant melanoma. Cancer Chemother Pharmacol. 1990;25(4):263-6. doi: 10.1007/BF00684883. PMID 2403853
- [Background] Bignami M, O'Driscoll M, Aquilina G, Karran P. Unmasking a killer: DNA O(6)-methylguanine and the cytotoxicity of methylating agents. Mutat Res. 2000 Apr;462(2-3):71-82. doi: 10.1016/s1383-5742(00)00016-8. PMID 10767619
- [Background] Lissoni P, Barni S, Tancini G, Ardizzoia A, Ricci G, Aldeghi R, Brivio F, Tisi E, Rovelli F, Rescaldani R, et al. A randomised study with subcutaneous low-dose interleukin 2 alone vs interleukin 2 plus the pineal neurohormone melatonin in advanced solid neoplasms other than renal cancer and melanoma. Br J Cancer. 1994 Jan;69(1):196-9. doi: 10.1038/bjc.1994.34. PMID 8286206
- [Background] Preuss I, Thust R, Kaina B. Protective effect of O6-methylguanine-DNA methyltransferase (MGMT) on the cytotoxic and recombinogenic activity of different antineoplastic drugs. Int J Cancer. 1996 Feb 8;65(4):506-12. doi: 10.1002/(SICI)1097-0215(19960208)65:43.0.CO;2-7. PMID 8621235
- [Background] Becker K, Gregel CM, Kaina B. The DNA repair protein O6-methylguanine-DNA methyltransferase protects against skin tumor formation induced by antineoplastic chloroethylnitrosourea. Cancer Res. 1997 Aug 15;57(16):3335-8. PMID 9269990
- [Background] Wibley JE, Pegg AE, Moody PC. Crystal structure of the human O(6)-alkylguanine-DNA alkyltransferase. Nucleic Acids Res. 2000 Jan 15;28(2):393-401. doi: 10.1093/nar/28.2.393. PMID 10606635
- [Background] Griffin RJ, Arris CE, Bleasdale C, Boyle FT, Calvert AH, Curtin NJ, Dalby C, Kanugula S, Lembicz NK, Newell DR, Pegg AE, Golding BT. Resistance-modifying agents. 8. Inhibition of O(6)-alkylguanine-DNA alkyltransferase by O(6)-alkenyl-, O(6)-cycloalkenyl-, and O(6)-(2-oxoalkyl)guanines and potentiation of temozolomide cytotoxicity in vitro by O(6)-(1-cyclopentenylmethyl)guanine. J Med Chem. 2000 Nov 2;43(22):4071-83. doi: 10.1021/jm000961o. PMID 11063604
- [Background] Daniels DS, Tainer JA. Conserved structural motifs governing the stoichiometric repair of alkylated DNA by O(6)-alkylguanine-DNA alkyltransferase. Mutat Res. 2000 Aug 30;460(3-4):151-63. doi: 10.1016/s0921-8777(00)00024-0. PMID 10946226
- [Background] Mineura K, Yanagisawa T, Watanabe K, Kowada M, Yasui N. Human brain tumor O(6)-methylguanine-DNA methyltransferase mRNA and its significance as an indicator of selective chloroethylnitrosourea chemotherapy. Int J Cancer. 1996 Oct 21;69(5):420-5. doi: 10.1002/(SICI)1097-0215(19961021)69:53.0.CO;2-6. PMID 8900378
- [Background] Alvino E, Pepponi R, Pagani E, Lacal PM, Nunziata C, Bonmassar E, D'Atri S. O(6)-benzylguanine enhances the in vitro immunotoxic activity of temozolomide on natural or antigen-dependent immunity. J Pharmacol Exp Ther. 1999 Dec;291(3):1292-300. PMID 10565854
- [Background] Davis BM, Roth JC, Liu L, Xu-Welliver M, Pegg AE, Gerson SL. Characterization of the P140K, PVP(138-140)MLK, and G156A O6-methylguanine-DNA methyltransferase mutants: implications for drug resistance gene therapy. Hum Gene Ther. 1999 Nov 20;10(17):2769-78. doi: 10.1089/10430349950016500. PMID 10584923
- [Background] Reese JS, Koc ON, Lee KM, Liu L, Allay JA, Phillips WP Jr, Gerson SL. Retroviral transduction of a mutant methylguanine DNA methyltransferase gene into human CD34 cells confers resistance to O6-benzylguanine plus 1,3-bis(2-chloroethyl)-1-nitrosourea. Proc Natl Acad Sci U S A. 1996 Nov 26;93(24):14088-93. doi: 10.1073/pnas.93.24.14088. PMID 8943065
- [Background] Mineura K, Fukuchi M, Kowada M, Terashima I, Kohda K. Differential inactivation of O6-methylguanine-DNA methyltransferase activity by O6-arylmethylguanines. Int J Cancer. 1995 Sep 27;63(1):148-51. doi: 10.1002/ijc.2910630126. PMID 7558444
- [Background] Bearzatto A, Szadkowski M, Macpherson P, Jiricny J, Karran P. Epigenetic regulation of the MGMT and hMSH6 DNA repair genes in cells resistant to methylating agents. Cancer Res. 2000 Jun 15;60(12):3262-70. PMID 10866320
- [Background] von Wronski MA, Brent TP. Effect of 5-azacytidine on expression of the human DNA repair enzyme O6-methylguanine-DNA methyltransferase. Carcinogenesis. 1994 Apr;15(4):577-82. doi: 10.1093/carcin/15.4.577. PMID 7511991
- [Background] Bhakat KK, Mitra S. Regulation of the human O(6)-methylguanine-DNA methyltransferase gene by transcriptional coactivators cAMP response element-binding protein-binding protein and p300. J Biol Chem. 2000 Nov 3;275(44):34197-204. doi: 10.1074/jbc.M005447200. PMID 10942771
- [Background] Esteller M, Garcia-Foncillas J, Andion E, Goodman SN, Hidalgo OF, Vanaclocha V, Baylin SB, Herman JG. Inactivation of the DNA-repair gene MGMT and the clinical response of gliomas to alkylating agents. N Engl J Med. 2000 Nov 9;343(19):1350-4. doi: 10.1056/NEJM200011093431901. Erratum In: N Engl J Med 2000 Dec 7;343(23):1740. PMID 11070098
- [Background] Slack A, Cervoni N, Pinard M, Szyf M. Feedback regulation of DNA methyltransferase gene expression by methylation. Eur J Biochem. 1999 Aug;264(1):191-9. doi: 10.1046/j.1432-1327.1999.00603.x. PMID 10447688